CLINICAL TRIAL: NCT05623553
Title: Evaluation of a Smartphone Based Diagnostic Tool to Assess Neonatal Jaundice in a Mexican Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Picterus AS (Industry)
Collaborators: Norwegian University of Science and Technology Faculty of Medicine and Health Sciences Department of Public Health and Nursing (Unknown); Hospital Materno- Infantil de Irapuato (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2018/1001
Record Dates: First submitted 2022-11-08; First posted 2022-11-21 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Jaundice, Neonatal
MeSH Terms: conditions — Jaundice, Neonatal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enable high qualitative estimation of bilirubin levels in the blood of new-borns (Experimental): There is only one arm in this study which is to enable high qualitative estimation of bilirubin levels in the blood of new-borns, independent of skin color, using Picterus JP.
  Interventions: Device: Picterus Jaundice Pro

INTERVENTIONS:
Device: Picterus Jaundice Pro — Use Picterus Jaundice Pro, a smartphone app that is used to take photo of the newborns skin, where the Picterus calibration card is place.
  Other Names: Picterus JP

SUMMARY:
This corss-sectional study aims to test the performance and accuracy of the Picterus JP screening device in newborns with different skin types.

DETAILED DESCRIPTION:
A descriptive cross-sectional study among 174 newborns was carried out at Hospital Materno-Infantil de Irapuato in Mexico during July and August 2018.

The Picterus Calibration Card will be placed on the chest of the newborn with the hole in the card placed over the infant's sternum. A validated smartphone with Picterus JP will be used to collect digital images..

ELIGIBILITY:
Inclusion Criteria:

* Healthy newborns with or without signs of jaundice
* Gestational age >35 weeks
* Age 0-14 days
* Birth weight > 1500 g.
* Parents acceptance of their children to participate in the study.
* Newborn needing a blood test

Exclusion Criteria:

* Newborns showing signs or with diagnosis of inborn diseases
* Newborn transferred to pediatric ward for any treatment
* Newborns who had received phototherapy.

Ages: 0 Days to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 174 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-07-11 (Actual); Study Completion 2018-08-08 (Actual)

PRIMARY OUTCOMES:
Enable high qualitative estimation of bilirubin levels in the blood of newborns using Picterus JP | 6 months
  Evaluate of smartphone-based diagnostic tool (Picterus JP) for neonatal jaundice in newborns.

SECONDARY OUTCOMES:
Correlation with TsB | 1-2 hours
  Demonstrate the correlation among the estimated levels of bilirubin obtained through a smartphone based diagnostic tool with bilirubin serum levels in a population of Mexican neonates.
Correlation with TcB | 5-10 minutes
  Demonstrate the correlation among the estimated levels of bilirubin obtained through a smartphone based diagnostic tool with those obtained using a transcutaneous bilirubinometer in a population of Mexican neonates.
Correlation with visual assessment | 5-10 minutes
  Demonstrate the correlation among the estimated levels of bilirubin obtained through a smartphone based diagnostic tool with those obtained using visual Kramer scale in a population of Mexican neonates.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Darj, Prof, MD, PhD, Principal Investigator — NTNU Faculty of Medicine and Health Sciences, Department of Public Health and Nursing
Locations (1):
- Hospital Materno- Infantil de Irapuato, Irapuato, Guanajuato, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Master thesis describing the study and its results — https://www.google.com/url?sa=t&rct=j&q=&esrc=s&source=web&cd=&cad=rja&uact=8&ved=2ahUKEwjw9pvJvpz7AhWGaMAKHVWXB3EQFnoECF0QAQ&url=https%3A%2F%2Fntnuopen.ntnu.no%2Fntnu-xmlui%2Fbitstream%2Fhandle%2F11250%2F2616837%2Fno.ntnu%253Ainspera%253A2379649.pdf%3Fsequence%3D1&usg=AOvVaw10PdE6VGVgBoTdKsQ-0AUs